CLINICAL TRIAL: NCT00002540
Title: Prostate, Lung, Colorectal, and Ovarian (PLCO) Cancer Screening Trial
Brief Title: Screening for Prostate Cancer in Older Patients (PLCO Screening Trial)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: NCI-2012-01755; NCI-2012-01755 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000078532; NCI-P93-0050; PLCO-1; PLCO-Prostate (Other: National Cancer Institute)
Record Dates: First submitted 1999-11-01; First posted 2004-03-26 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Restraint, Physical; Nutrition Surveys; Independent Medical Evaluation

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- Control (No Intervention): Participants receive standard medical care. Participants complete a DHQ at baseline.
- Prostate Screening (Active Comparator): Participants undergo blood sample collection for PSA analysis at baseline and annually for 5 years. Serum that is not used in the study will be stored in an NCI biorepository. Participants also undergo a DRE at baseline and annually for 3 years. Participants complete a DQX at baseline and DHQ at year 3. An ADU (previously referred to as the PSH questionnaire) is mailed to each participant annually for 13 years to identify all prevalent and incident prostate cancers as all deaths that occur among both screened and control subjects during the trial.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Medical Examination Assessment; Other: Screening Questionnaire Administration

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
  Arms: Prostate Screening
Procedure: Medical Examination Assessment — Undergo DRE
  Other Names: Exam; Examination; Health Assessment; Health Examination; Health Status Assessment; Medical Assessment; Medical Exam; Medical Inspection
  Arms: Prostate Screening
Other: Screening Questionnaire Administration — Undergo questionnaire assessments
  Arms: Prostate Screening

SUMMARY:
This clinical trial studies whether screening methods used to diagnose cancer of the prostate, lung, colon, rectum, or ovaries can reduce deaths from these cancers. Screening tests may help doctors find cancer cells early and plan better treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine whether screening with digital rectal examination (DRE) plus serum prostate-specific antigen (PSA) can reduce mortality from prostate cancer in men aged 55-74 at entry.

SECONDARY OBJECTIVES:

I. To assess screening variables, other than mortality, for each of the interventions including sensitivity, specificity, and positive predictive value.

II. To assess the incidence, stage, and survival of cancer cases. III. To investigate the mortality predictive value of biologic and/or prognostic characterizations of tumor tissue as intermediate endpoints.

IV. To conduct biomolecular and genetic research into factors associated with cancer carcinogenesis and promotion, as well as the early detection of these factors.

OUTLINE: Participants in the overall PLCO study are stratified by screening center, gender, and age (55-59 vs 60-64 vs 65-69 vs 70-74). Participants are randomized to 1 of 2 arms (control vs screening).

ARM I (Control): Participants receive standard medical care. Participants complete a Diet History Questionnaire (DHQ) at baseline.

ARM II (Prostate Screening): Participants undergo blood sample collection for PSA analysis at baseline and annually for 5 years. Serum that is not used in the study will be stored in an NCI biorepository. Participants also undergo a DRE at baseline and annually for 3 years. A scheduling and tracking procedure is implemented to ensure regular attendance at repeat screens for participants screened negative or for those who are designated suspicious or positive at screening but for whom subsequent diagnostic procedures do not reveal prostate cancer (follow-up diagnostic procedures are through their own medical care environment). Participants diagnosed with prostate cancer via a screening test are referred for treatment in accordance with current accepted practice for appropriate stage of disease, patient age, and medical condition; a procedure is provided for contact with qualified medical personnel to insure appropriate therapy.

Participants complete a Dietary Questionnaire (DQX) at baseline and DHQ at year 3. An Annual Study Update (ADU) (previously referred to as the Periodic Survey of Health [PSH] questionnaire) is mailed to each participant annually for 13 years to identify all prevalent and incident prostate cancers as all deaths that occur among both screened and control subjects during the trial.

After completion of screening, participants are followed up for at least 13 years.

ELIGIBILITY:
Exclusion Criteria:

* Men who at the time of randomization are less than 55 or greater than or equal to 75 years of age
* Individuals undergoing treatment for cancer at this time, excluding basal-cell and squamous-cell skin cancer
* Individuals with known prior cancer of the colon, rectum, lung, prostate

  * This includes primary or metastatic PLCO cancers
* Individuals with previous surgical removal of the entire colon, one lung, or the entire prostate
* Individuals who are participating in another cancer screening or cancer primary prevention trial
* Males who have taken Proscar/Propecia/finasteride in the past 6 months

  * NOTE: Individuals who are already enrolled in the trial when their physician prescribes finasteride are not prevented from taking this medication. As a result, these participants will continue to be screened and followed just as those participants who are not on finasteride.
  * NOTE: Men who are taking Tamoxifen are not excluded from any part of the PLCO Screening Trial.
* Individuals who are unwilling or unable to sign the informed consent form
* Males who have had more than one PSA blood test in the past three years
* Individuals who have had a colonoscopy, sigmoidoscopy, or barium enema in the past three years

Ages: 55 Years to 74 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76685 (Actual)
Dates: Start 1993-11-16 (Actual); Primary Completion 2012-05-21 (Actual); Study Completion 2026-03-25 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Christine D Berg, Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Malcomson FC, Shams-White MM, Reedy J, Huang WY, Moore SC, Loftfield E. Adherence to the 2018 World Cancer Research Fund/American Institute for Cancer Research Cancer Prevention Recommendations and risk of lifestyle-related cancers in the prostate, lung, colorectal, and ovarian cancer screening trial. BJC Rep. 2025 Nov 19;3(1):81. doi: 10.1038/s44276-025-00195-6. PMID 41261199
- [Derived] Fan Z, Zhang Y, Yao Q, Liu X, Duan H, Liu Y, Sheng C, Lyu Z, Yang L, Song F, Huang Y, Song F. Effects of joint screening for prostate, lung, colorectal, and ovarian cancer - results from a controlled trial. Front Oncol. 2024 Apr 29;14:1322044. doi: 10.3389/fonc.2024.1322044. eCollection 2024. PMID 38741776
- [Derived] Jiang Y, Xie Q, Chen R. Breast Cancer Incidence and Mortality in Relation to Hormone Replacement Therapy Use Among Postmenopausal Women: Results From a Prospective Cohort Study. Clin Breast Cancer. 2022 Feb;22(2):e206-e213. doi: 10.1016/j.clbc.2021.06.010. Epub 2021 Jun 26. PMID 34548240
- [Derived] Pinsky PF, Durham D, Strassels S. Opioid and Other Medication Use and General Health Status in a Cohort of Older Adults. Gerontology. 2021;67(5):554-562. doi: 10.1159/000513731. Epub 2021 Mar 10. PMID 33691305
- [Derived] Wang K, Wu Q, Li Z, Reger MK, Xiong Y, Zhong G, Li Q, Zhang X, Li H, Foukakis T, Xiang T, Zhang J, Ren G. Vitamin K intake and breast cancer incidence and death: results from a prospective cohort study. Clin Nutr. 2021 May;40(5):3370-3378. doi: 10.1016/j.clnu.2020.11.009. Epub 2020 Nov 16. PMID 33277073
- [Derived] Pinsky PF, Miller EA, Zhu CS, Prorok PC. Overall mortality in men and women in the randomized Prostate, Lung, Colorectal, and Ovarian Cancer Screening Trial. J Med Screen. 2019 Sep;26(3):127-134. doi: 10.1177/0969141319839097. Epub 2019 Apr 3. No abstract available. PMID 30943843
- [Derived] Pierre-Victor D, Pinsky PF. Association of Nonadherence to Cancer Screening Examinations With Mortality From Unrelated Causes: A Secondary Analysis of the PLCO Cancer Screening Trial. JAMA Intern Med. 2019 Feb 1;179(2):196-203. doi: 10.1001/jamainternmed.2018.5982. PMID 30592477
- [Derived] Miller EA, Pinsky PF, Schoen RE, Prorok PC, Church TR. Effect of flexible sigmoidoscopy screening on colorectal cancer incidence and mortality: long-term follow-up of the randomised US PLCO cancer screening trial. Lancet Gastroenterol Hepatol. 2019 Feb;4(2):101-110. doi: 10.1016/S2468-1253(18)30358-3. Epub 2018 Nov 29. PMID 30502933
- [Derived] Click B, Pinsky PF, Hickey T, Doroudi M, Schoen RE. Association of Colonoscopy Adenoma Findings With Long-term Colorectal Cancer Incidence. JAMA. 2018 May 15;319(19):2021-2031. doi: 10.1001/jama.2018.5809. PMID 29800214
- [Derived] Schoen RE, Razzak A, Yu KJ, Berndt SI, Firl K, Riley TL, Pinsky PF. Incidence and mortality of colorectal cancer in individuals with a family history of colorectal cancer. Gastroenterology. 2015 Nov;149(6):1438-1445.e1. doi: 10.1053/j.gastro.2015.07.055. Epub 2015 Aug 5. PMID 26255045
- [Derived] Guertin KA, Loftfield E, Boca SM, Sampson JN, Moore SC, Xiao Q, Huang WY, Xiong X, Freedman ND, Cross AJ, Sinha R. Serum biomarkers of habitual coffee consumption may provide insight into the mechanism underlying the association between coffee consumption and colorectal cancer. Am J Clin Nutr. 2015 May;101(5):1000-11. doi: 10.3945/ajcn.114.096099. Epub 2015 Mar 11. PMID 25762808
- [Derived] Kvale PA, Johnson CC, Tammemagi M, Marcus PM, Zylak CJ, Spizarny DL, Hocking W, Oken M, Commins J, Ragard L, Hu P, Berg C, Prorok P. Interval lung cancers not detected on screening chest X-rays: How are they different? Lung Cancer. 2014 Oct;86(1):41-6. doi: 10.1016/j.lungcan.2014.07.013. Epub 2014 Jul 24. PMID 25123333
- [Derived] Guertin KA, Moore SC, Sampson JN, Huang WY, Xiao Q, Stolzenberg-Solomon RZ, Sinha R, Cross AJ. Metabolomics in nutritional epidemiology: identifying metabolites associated with diet and quantifying their potential to uncover diet-disease relations in populations. Am J Clin Nutr. 2014 Jul;100(1):208-17. doi: 10.3945/ajcn.113.078758. Epub 2014 Apr 16. PMID 24740205
- [Derived] Major JM, Yu K, Weinstein SJ, Berndt SI, Hyland PL, Yeager M, Chanock S, Albanes D. Genetic variants reflecting higher vitamin e status in men are associated with reduced risk of prostate cancer. J Nutr. 2014 May;144(5):729-33. doi: 10.3945/jn.113.189928. Epub 2014 Mar 12. PMID 24623848
- [Derived] Hocking WG, Tammemagi MC, Commins J, Oken MM, Kvale PA, Hu P, Ragard LR, Riley TL, Pinsky P, Beck TM, Prorok PC. Diagnostic evaluation following a positive lung screening chest radiograph in the Prostate, Lung, Colorectal, Ovarian (PLCO) Cancer Screening Trial. Lung Cancer. 2013 Nov;82(2):238-44. doi: 10.1016/j.lungcan.2013.07.017. Epub 2013 Aug 7. PMID 23993734
- [Derived] Rogal SS, Pinsky PF, Schoen RE. Relationship between detection of adenomas by flexible sigmoidoscopy and interval distal colorectal cancer. Clin Gastroenterol Hepatol. 2013 Jan;11(1):73-8. doi: 10.1016/j.cgh.2012.08.002. Epub 2012 Aug 16. PMID 22902761
- [Derived] Schoen RE, Pinsky PF, Weissfeld JL, Yokochi LA, Church T, Laiyemo AO, Bresalier R, Andriole GL, Buys SS, Crawford ED, Fouad MN, Isaacs C, Johnson CC, Reding DJ, O'Brien B, Carrick DM, Wright P, Riley TL, Purdue MP, Izmirlian G, Kramer BS, Miller AB, Gohagan JK, Prorok PC, Berg CD; PLCO Project Team. Colorectal-cancer incidence and mortality with screening flexible sigmoidoscopy. N Engl J Med. 2012 Jun 21;366(25):2345-57. doi: 10.1056/NEJMoa1114635. Epub 2012 May 21. PMID 22612596
- [Derived] Oken MM, Hocking WG, Kvale PA, Andriole GL, Buys SS, Church TR, Crawford ED, Fouad MN, Isaacs C, Reding DJ, Weissfeld JL, Yokochi LA, O'Brien B, Ragard LR, Rathmell JM, Riley TL, Wright P, Caparaso N, Hu P, Izmirlian G, Pinsky PF, Prorok PC, Kramer BS, Miller AB, Gohagan JK, Berg CD; PLCO Project Team. Screening by chest radiograph and lung cancer mortality: the Prostate, Lung, Colorectal, and Ovarian (PLCO) randomized trial. JAMA. 2011 Nov 2;306(17):1865-73. doi: 10.1001/jama.2011.1591. Epub 2011 Oct 26. PMID 22031728
- [Derived] Buys SS, Partridge E, Black A, Johnson CC, Lamerato L, Isaacs C, Reding DJ, Greenlee RT, Yokochi LA, Kessel B, Crawford ED, Church TR, Andriole GL, Weissfeld JL, Fouad MN, Chia D, O'Brien B, Ragard LR, Clapp JD, Rathmell JM, Riley TL, Hartge P, Pinsky PF, Zhu CS, Izmirlian G, Kramer BS, Miller AB, Xu JL, Prorok PC, Gohagan JK, Berg CD; PLCO Project Team. Effect of screening on ovarian cancer mortality: the Prostate, Lung, Colorectal and Ovarian (PLCO) Cancer Screening Randomized Controlled Trial. JAMA. 2011 Jun 8;305(22):2295-303. doi: 10.1001/jama.2011.766. PMID 21642681
- [Derived] Berg CD. The Prostate, Lung, Colorectal and Ovarian Cancer Screening Trial: the prostate cancer screening results in context. Acta Oncol. 2011 Jun;50 Suppl 1:12-7. doi: 10.3109/0284186X.2010.531283. PMID 21604935
- [Derived] Pinsky PF, Blacka A, Kramer BS, Miller A, Prorok PC, Berg C. Assessing contamination and compliance in the prostate component of the Prostate, Lung, Colorectal, and Ovarian (PLCO) Cancer Screening Trial. Clin Trials. 2010 Aug;7(4):303-11. doi: 10.1177/1740774510374091. Epub 2010 Jun 22. PMID 20571134
- [Derived] Troy JD, Hartge P, Weissfeld JL, Oken MM, Colditz GA, Mechanic LE, Morton LM. Associations between anthropometry, cigarette smoking, alcohol consumption, and non-Hodgkin lymphoma in the Prostate, Lung, Colorectal, and Ovarian Cancer Screening Trial. Am J Epidemiol. 2010 Jun 15;171(12):1270-81. doi: 10.1093/aje/kwq085. Epub 2010 May 21. PMID 20494998
- [Derived] Croswell JM, Kramer BS, Kreimer AR, Prorok PC, Xu JL, Baker SG, Fagerstrom R, Riley TL, Clapp JD, Berg CD, Gohagan JK, Andriole GL, Chia D, Church TR, Crawford ED, Fouad MN, Gelmann EP, Lamerato L, Reding DJ, Schoen RE. Cumulative incidence of false-positive results in repeated, multimodal cancer screening. Ann Fam Med. 2009 May-Jun;7(3):212-22. doi: 10.1370/afm.942. PMID 19433838
- [Derived] Tammemagi MC, Freedman MT, Pinsky PF, Oken MM, Hu P, Riley TL, Ragard LR, Berg CD, Prorok PC. Prediction of true positive lung cancers in individuals with abnormal suspicious chest radiographs: a prostate, lung, colorectal, and ovarian cancer screening trial study. J Thorac Oncol. 2009 Jun;4(6):710-21. doi: 10.1097/JTO.0b013e31819e77ce. PMID 19404219
- [Derived] Partridge E, Kreimer AR, Greenlee RT, Williams C, Xu JL, Church TR, Kessel B, Johnson CC, Weissfeld JL, Isaacs C, Andriole GL, Ogden S, Ragard LR, Buys SS; PLCO Project Team. Results from four rounds of ovarian cancer screening in a randomized trial. Obstet Gynecol. 2009 Apr;113(4):775-782. doi: 10.1097/AOG.0b013e31819cda77. PMID 19305319
- [Derived] Andriole GL, Crawford ED, Grubb RL 3rd, Buys SS, Chia D, Church TR, Fouad MN, Gelmann EP, Kvale PA, Reding DJ, Weissfeld JL, Yokochi LA, O'Brien B, Clapp JD, Rathmell JM, Riley TL, Hayes RB, Kramer BS, Izmirlian G, Miller AB, Pinsky PF, Prorok PC, Gohagan JK, Berg CD; PLCO Project Team. Mortality results from a randomized prostate-cancer screening trial. N Engl J Med. 2009 Mar 26;360(13):1310-9. doi: 10.1056/NEJMoa0810696. Epub 2009 Mar 18. PMID 19297565
- [Derived] Lacey JV Jr, Kreimer AR, Buys SS, Marcus PM, Chang SC, Leitzmann MF, Hoover RN, Prorok PC, Berg CD, Hartge P; Prostate, Lung, Colorectal and Ovarian (PLCO) Cancer Screening Trial Project Team. Breast cancer epidemiology according to recognized breast cancer risk factors in the Prostate, Lung, Colorectal and Ovarian (PLCO) Cancer Screening Trial Cohort. BMC Cancer. 2009 Mar 17;9:84. doi: 10.1186/1471-2407-9-84. PMID 19292893
- [Derived] Tammemagi CM, Freedman MT, Church TR, Oken MM, Hocking WG, Kvale PA, Hu P, Riley TL, Ragard LR, Prorok PC, Berg CD. Factors associated with human small aggressive non small cell lung cancer. Cancer Epidemiol Biomarkers Prev. 2007 Oct;16(10):2082-9. doi: 10.1158/1055-9965.EPI-07-0251. PMID 17932357
- [Derived] Lacey JV Jr, Greene MH, Buys SS, Reding D, Riley TL, Berg CD, Fagerstrom RM, Hartge P. Ovarian cancer screening in women with a family history of breast or ovarian cancer. Obstet Gynecol. 2006 Nov;108(5):1176-84. doi: 10.1097/01.AOG.0000239105.39149.d8. PMID 17077240

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between November 1993 and July 2001 at 10 study centers. Recruitment was done for all four outcomes of the study (prostate, lung, colorectal and ovarian).
Pre-assignment Details: Participants signed a study informed consent prior to being randomized to a study arm.
Groups:
- Control: Participants receive standard medical care.
- Prostate Screening: Participants undergo blood sample collection for prostate specific antigen (PSA) analysis at baseline and annually for 5 years. Participants also undergo a digital rectal examination (DRE) at baseline and annually for 3 years.
Period: Overall Study
Arm/Group | Control | Prostate Screening
Started | 38345 | 38340
Completed | 37544 | 35876
Not Completed | 801 | 2464
Not completed — Cancer Before Rand. (Prostate Screening) | 0 | 25
Not completed — Died Before Randomization | 2 | 6
Not completed — Died Before ASU (Control) | 202 | 0
Not completed — Refused ASU (Control) | 597 | 0
Not completed — Refused Screen (Prostate Screening) | 0 | 2433

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Prostate Screening | Total
Number analyzed (Participants) | 38345 | 38340 | 76685
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24390 | 24400 | 48790
  >=65 years | 13955 | 13940 | 27895
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.7 (5.3) | 62.7 (5.3) | 62.7 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 38345 | 38340 | 76685
Region of Enrollment [Number; unit: participants]
  United States | 38345 | 38340 | 76685

OUTCOME MEASURES:

1. Primary Outcome: Prostate Cancer Deaths
Description: Prostate cancer deaths confirmed in participants by a death review committee if available, otherwise by death certificate.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 12.0 years.
Population: All male participants randomized were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Arm/Group | Control | Prostate Screening
Number analyzed (Participants) | 38345 | 38340
Participants | 145 | 158
Statistical Analysis 1: Comparison: Control vs Prostate Screening; Test type: Superiority or Other; Poisson regression — Two-sided. Not adjusted for multiple comparisons. A-priori threshold for significance 0.05; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.87 to 1.36]

2. Secondary Outcome: Deaths From All Causes
Description: Deaths from all causes were compared between the prostate cancer screening arm and the usual care arm.
Time Frame: Events through 13 years of follow-up or through December 31, 2009.
Population: All male participants were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Arm/Group | Control | Prostate Screening
Number analyzed (Participants) | 38345 | 38340
Participants | 7089 | 6855

3. Secondary Outcome: Death Rates From All Causes
Description: Deaths from all causes were compared between the prostate cancer screening arm and the usual care arm. Rate is the number of deaths divided by person years of follow-up in the study.
Time Frame: Events through 13 years of follow-up or through December 31, 2009.
Population: All male participants were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Deaths per 10,000 PY
Arm/Group | Control | Prostate Screening
Number analyzed (Participants) | 38345 | 38340
Deaths per 10,000 PY | 166.6 | 160.5
Statistical Analysis 1: Comparison: Control vs Prostate Screening; Test type: Superiority or Other; Poisson regression; Two-sided. Not adjusted for multiple comparisons. A-priori threshold for significance 0.05; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.93 to 1.00]

4. Secondary Outcome: Prostate Cancer Incidence
Description: Prostate cancer diagnoses confirmed by medical record abstraction. Incidence rate (cumulative) defined as prostate cancer diagnoses divided by person years at risk for prostate cancer.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 12.0 years.
Population: All male participants randomized were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Participants
Arm/Group | Control | Prostate Screening
Number analyzed (Participants) | 38345 | 38340
Participants | 3815 | 4250

5. Secondary Outcome: Prostate Cancer Incidence Rates
Description: as for outcome 4
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 12.0 years.
Population: All male participants randomized were analyzed. An intention-to-treat analysis was performed.
Measure: Number; unit: Diagnoses per 10,000 PY
Arm/Group | Control | Prostate Screening
Number analyzed (Participants) | 38345 | 38340
Diagnoses per 10,000 PY | 97.1 | 108.4
Statistical Analysis 1: Comparison: Control vs Prostate Screening; Test type: Superiority or Other; Poisson regression; Two-sided. Not adjusted for multiple comparisons. A-priori threshold for significance 0.05; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [1.07 to 1.17]

6. Secondary Outcome: Complications of Diagnostic Evaluation (DE) Following a Positive Screening Test
Description: Number of positive screens with complications
Time Frame: One year from screening examination
Population: The units analyzed were positive screening exams with documented diagnostic follow-up. If a participant received 3 positive screens with documented follow-up after each one, he would be counted 3 times in the number of units analyzed.
Measure: Number; unit: Positive screens w/ complications
Units Other Than Participants: Positive Screens with Follow-up
Arm/Group | Prostate Screening
Number analyzed (Participants) | 10642
Number analyzed (Positive Screens with Follow-up) | 22269
Positive screens w/ complications
  When DE Led to Prostate Cancer Diagnosis | 901
  When DE Did Not Lead to Prostate Cancer Diagnosis | 124

7. Secondary Outcome: T0 (Baseline) PSA Screening Results
Description: Prostate-Specific Antigen (PSA) result.
Time Frame: T0 (at study entry)
Population: All males in the Prostate Screening arm who had a PSA screen at T0 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Prostate Screening
Number analyzed (Participants) | 34247
Participants
  Negative (<=4 ng/mL) | 31507
  Positive (> 4 ng/mL) | 2718
  Inadequate screen | 22

8. Secondary Outcome: T0 (Baseline) DRE Screening Results
Description: Digital Rectal Examination (DRE) result.
Time Frame: T0 (at study entry)
Population: All males in the Prostate Screening arm who had a DRE screen at T0 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Prostate Screening
Number analyzed (Participants) | 34129
Participants
  Negative | 30456
  Positive | 2481
  Inadequate screen | 1192

9. Secondary Outcome: T1 PSA Screening Results
Description: Prostate-Specific Antigen (PSA) result.
Time Frame: T1 (one year after entry)
Population: All males in the Prostate Screening arm who had a PSA screen at T1 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Prostate Screening
Number analyzed (Participants) | 32688
Participants
  Negative (<=4 ng/mL) | 30159
  Positive (> 4 ng/mL) | 2502
  Inadequate screen | 27

10. Secondary Outcome: T1 DRE Screening Results
Description: Digital Rectal Examination (DRE) result.
Time Frame: T1 (one year after entry)
Population: All males in the Prostate Screening arm who had a DRE screen at T1 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Prostate Screening
Number analyzed (Participants) | 32448
Participants
  Negative | 29311
  Positive | 2237
  Inadequate screen | 900

11. Secondary Outcome: T2 PSA Screening Results
Description: Prostate-Specific Antigen (PSA) result.
Time Frame: T2 (two years after entry)
Population: All males in the Prostate Screening arm who had a PSA screen at T2 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Prostate Screening
Number analyzed (Participants) | 31691
Participants
  Negative | 29063
  Positive (> 4 ng/mL) | 2593
  Inadequate screen | 35

12. Secondary Outcome: T2 DRE Screening Results
Description: Digital Rectal Examination (DRE) results
Time Frame: T2 (two years after entry)
Population: All males in the Prostate Screening arm who had a DRE screen at T2 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Prostate Screening
Number analyzed (Participants) | 31451
Participants
  Negative | 28391
  Positive | 2327
  Inadequate screen | 733

13. Secondary Outcome: T3 PSA Screening Results
Description: Prostate-Specific Antigen (PSA) result
Time Frame: T3 (three years after entry)
Population: All males in the Prostate Screening arm who had a PSA screen at T3 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Prostate Screening
Number analyzed (Participants) | 30533
Participants
  Negative (<=4 ng/mL) | 27814
  Positive (> 4 ng/mL) | 2676
  Inadequate screen | 43

14. Secondary Outcome: T3 DRE Screening Results
Description: Digital Rectal examination (DRE) result
Time Frame: T3 (three years after entry)
Population: All males in the Prostate Screening arm who had a DRE screen at T3 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Prostate Screening
Number analyzed (Participants) | 30244
Participants
  Negative | 27179
  Positive | 2317
  Inadequate screen | 748

15. Primary Outcome: Prostate Cancer Death Rates
Description: Prostate cancer deaths confirmed in participants by a death review committee if available, otherwise by death certificate. Rate is the number of deaths divided by person years of follow-up in the study.
Time Frame: Events through 13 years of follow-up or through December 31, 2009; median follow-up 12.0 years.
Measure: Number; unit: Deaths per 10,000 PY
Arm/Group | Control | Prostate Screening
Number analyzed (Participants) | 38345 | 38340
Deaths per 10,000 PY | 3.4 | 3.7
Statistical Analysis 1: Comparison: Control vs Prostate Screening; Test type: Superiority or Other; Poisson regression; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.87 to 1.36]

16. Secondary Outcome: T4 PSA Screening Result
Description: Prostate-Specific Antigen (PSA) result
Time Frame: T4 (four years after entry)
Population: All males in the Prostate Screening arm who had a PSA screen at T4 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Prostate Screening
Number analyzed (Participants) | 22170
Participants
  Negative (<=4 ng/mL) | 20362
  Positive (> 4 ng/mL) | 1796
  Inadequate screen | 12

17. Secondary Outcome: T5 PSA Screening Results
Description: Prostate-Specific Antigen (PSA) result.
Time Frame: T5 (five years after entry)
Population: All males in the Prostate Screening arm who had a PSA screen at T5 were analyzed.
Measure: Number; unit: Participants
Arm/Group | Prostate Screening
Number analyzed (Participants) | 25951
Participants
  Negative (<=4 ng/mL) | 23560
  Positive (> 4 ng/mL) | 2377
  Inadequate screen | 14

ADVERSE EVENTS:
Time Frame: During each annual screening visit.
Description: These events are solely those prompted by the screening examination.
Arm/Group | Prostate Screening
Serious Adverse Events (participants affected / at risk) | 0/38340
Other Adverse Events (participants affected / at risk) | 546/38340
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prostate Screening (N=38340)
Anxiety (General disorders) | 1 (1)
Bleeding (General disorders) | 3 (3)
Dizzy (General disorders) | 101 (108)
Fainted (General disorders) | 58 (59)
Inflammation (General disorders) | 2 (2)
Nausea (General disorders) | 1 (1)
Pain (General disorders) | 11 (11)
Bruising (General disorders) | 182 (183)
Hematoma (General disorders) | 187 (190)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less